CLINICAL TRIAL: NCT01036035
Title: Effects of THVD-201 on Pharmacokinetics and Pharmacodynamics of Tolterodine in Healthy Subjects
Brief Title: Effects of Novel Combinations of Tolterodine/Pilocarpine on Pharmacokinetics (PK) and Pharmacodynamics (PD) of Tolterodine in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: TheraVida, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: THVD-201-001
Record Dates: First submitted 2009-12-16; First posted 2009-12-21 (Estimated); Last update posted 2015-12-30 (Estimated); Status verified 2015-12

CONDITIONS: Incontinence
Keywords: Tolterodine; Over active Bladder (OAB); Incontinence
MeSH Terms: interventions — Tolterodine Tartrate; Pilocarpine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Treatment B (Active Comparator): Study drug
  Interventions: Drug: Pilocarpine
- Treatment D (Active Comparator): Study drug
  Interventions: Drug: THVD-201
- Treatment E (Placebo Comparator): Placebo
  Interventions: Drug: placebo capsule
- Treatment A (Active Comparator): Study Drug
  Interventions: Drug: Tolterodine
- Treatment C (Active Comparator): Study Drug
  Interventions: Drug: THVD-201

INTERVENTIONS:
Drug: Tolterodine — Comparison of different dosages of drug
  Arms: Treatment A
Drug: Pilocarpine — Comparison of different dosages of drug
  Arms: Treatment B
Drug: THVD-201 — Comparison of different dosages of drug
  Arms: Treatment C
Drug: THVD-201 — Comparison of different dosages of drug
  Arms: Treatment D
Drug: placebo capsule — Comparison of different dosages of drug
  Arms: Treatment E

SUMMARY:
THVD-201 is a novel combination of a muscarinic antagonist (tolterodine) and a muscarinic agonist (pilocarpine).

DETAILED DESCRIPTION:
Because of the limitations of taking two medications separated by a period of time to minimise these adverse events, two novel formulations were developed to improve compliance and ease of administration. This study will evaluate these formulations in terms of their pharmacokinetic profiles and effects on SSF. In addition, the effects of this combination and its entities on urine frequency and safety/tolerability will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Healthy males, 18 - 45 years of age.
* BMI 20-30 m2.

Exclusion Criteria:

* Subjects who have a history of sensitivity to antimuscarinic or muscarinic agents or related derivatives.
* Clinically significant ECG, vital signs and clinical laboratory indices.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2009-09; Primary Completion 2010-03 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Reductions in stimulated salivary flow (SSF) | From Baseline

SECONDARY OUTCOMES:
Determine the pharmacokinetics of tolterodine and the agonist. | From Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Joanne Marjason, Principal Investigator — Queensland Institute for Medical Research